CLINICAL TRIAL: NCT03334552
Title: Identification of Broadly HIV-1 Neutralizing Antibodies (bNAb) in HIV-infected Patients in Mbeya, Tanzania.
Acronym: bNAb
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Michael Hoelscher (Other)
Collaborators: National Institute for Medical Research - Mbeya Medical Research Centre (NIMR-MMRC) (Unknown); University Clinic of Cologne, Department of Internal Medicine, Center for Molecular Medicine Cologne (CMMC) (Unknown); Max von Pettenkofer-Institute of the University of Munich (LMU), Department of Virology (Unknown)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Professor Dr., Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Other Study IDs: LMU-IMPH-bNAb
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In natural HIV disease, a small fraction (1-2%) of infected individuals develops exceptionally high titres of HIV-1 neutralizing serum activity. Antibodies isolated from these individuals have been shown to be highly active against a broad range of different HIV strains and are therefore called broadly neutralizing antibodies (bNAbs). These antibodies are in fact able to prevent (S)HIV infection in animal models and therefore of great interest for the development of an HIV vaccine. Information of neutralizing antibodies in patients from Africa is still scarce and would be of great value in the development of adapted HIV vaccine strategies in these regions. This study aims to investigate African HIV-infected individuals, who have developed neutralizing antibodies using highly specialized laboratory methodologies.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and informed consent
2. ≥18 years of age
3. Documented HIV infection.
4. Willing to consent to active tracing including home tracing

Exclusion Criteria:

1. Deficiency, rendering it difficult, if not impossible, to take part in the study or understand the information provided. This includes alcoholism, drug dependency as well as psychiatric illnesses, suicidal tendencies or any other inability.
2. Prisoners
3. If within the discretion of the investigator study participation would possibly add not acceptable risk or burden to patient (e.g. significant health deficiencies, social harm)
4. Unlikely to comply with protocol as judged by the principal investigator or his designate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult HIV-infected, preferentially ART-naïve patients within the Mbeya region. The prevalence of elite neutralizers is expected to be 1-2% from the overall population. The study therefore targets to recruit 500 subjects in order to identify at least 5 elite neutralizers, which will be subjected to further in depth antibody characterization.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Broadly HIV-1 neutralizing antibodies (bNAb) | December 31, 2018
  identify HIV-infected patients which exhibit exceptional HIV-1 neutralizing activity (so called elite neutralizer) and to perform in those patients in depth characterization including:
  * Detailed analysis of anti-HIV antibody response using single B cell analyis
  * Isolation of broadly neutralizing anti-HIV antibodies
  * Testing of in vitro neutralizing activity and binding properties of newly identified bNAbs
  * Analysis of the antiviral activity and in vivo characteristics of broadly neutralizing antibodies using a HIV-1-infected humanized mouse model

SECONDARY OUTCOMES:
To characterize HIV subtypes in elite neutralizer and optionally in non-neutralizer | December 31, 2018
To characterize demographic and HIV status related factors associated with elite neutralizers and non-neutralizers | December 31, 2018
To optionally investigate the proportion of patients with transmitted drug mutations (genotypic drug resistance) | December 31, 2018

CONTACTS AND LOCATIONS:
Overall Officials: Arne Kroidl, Dr., Study Chair — Medical Center of the University of Munich, Division of Infectious Diseases and Tropical Medicine, Germany; Wiston William, Dr., Principal Investigator — NIMR-Mbeya Medical Research Center (MMRC), Tazania
Locations (1):
- NIMR-Mbeya Medical Research Center (MMRC), Mbeya, Tanzania